CLINICAL TRIAL: NCT07394452
Title: A Phase 1 Clinical Trial to Evaluate the Safety, Tolerability, and Pharmacokinetics of TJ0113 Capsules Administered Orally as Single Dose, Multiple Doses, and Doses in the Fed State in Healthy Subjects
Brief Title: Single Ascending Dose Study(SAD),Multiple Ascending Dose Study(MAD) , High-fat Diet Study (FE) of TJ0113 Capsules in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hangzhou PhecdaMed Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TJJS01-001
Record Dates: First submitted 2026-01-26; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (13):
- Single Ascending Dose (SAD): 80 mg (Experimental): Participants will receive single oral administration of 80 mg TJ0113.
  Interventions: Drug: TJ0113 Capsules
- Single Ascending Dose (SAD): 160 mg (Experimental): Participants will receive single oral administration of 160 mg TJ0113.
  Interventions: Drug: TJ0113 Capsules
- Single Ascending Dose (SAD): 260 mg (Experimental): Participants will receive single oral administration of 260 mg TJ0113.
  Interventions: Drug: TJ0113 Capsules
- Single Ascending Dose (SAD): 400 mg (Experimental): Participants will receive single oral administration of 400 mg TJ0113.
  Interventions: Drug: TJ0113 Capsules
- Single Ascending Dose (SAD): 540 mg (Experimental): Participants will receive single oral administration of 540 mg TJ0113.
  Interventions: Drug: TJ0113 Capsules
- Single Ascending Dose (SAD): 720 mg (Experimental): Participants will receive single oral administration of 720 mg TJ0113.
  Interventions: Drug: TJ0113 Capsules
- Single Ascending Dose (SAD): placebo (Placebo Comparator): Participants will receive single oral administration of Placebo.
  Interventions: Other: Placebo
- Multiple Ascending Dose (MAD): 200 mg QD (Experimental): Participants will receive oral administration of 200 mg TJ0113 once daily for 7 days
  Interventions: Drug: TJ0113 Capsules
- Multiple Ascending Dose (MAD): 400 mg QD (Experimental): Participants will receive oral administration of 400 mg TJ0113 once daily for 7 days
  Interventions: Drug: TJ0113 Capsules
- Multiple Ascending Dose (MAD): 300 mg BID (Experimental): Participants will receive oral administration of 300 mg TJ0113 twice daily for 7 days
  Interventions: Drug: TJ0113 Capsules
- Multiple Ascending Dose (MAD): placebo (Placebo Comparator): Participants will receive oral administration of placebo for 7 days
  Interventions: Other: Placebo
- Food Effect: 200 mg C1: fasting-fed (Experimental): Group C1 received oral administration of 200 mg TJ0113 once in a fasting state during the first cycle and received oral administration of 200 mg TJ0113 once in a fed state during the second cycle. The two cycles were separated by a 7-day washout period.
  Interventions: Drug: TJ0113 Capsules
- Food Effect: 200 mg C2: fed-fasting (Experimental): Group C2 received oral administration of 200 mg TJ0113 once in a fed state during the first cycle and received oral administration of 200 mg TJ0113 once in a fasting state during the second cycle. The two cycles were separated by a 7-day washout period.
  Interventions: Drug: TJ0113 Capsules

INTERVENTIONS:
Drug: TJ0113 Capsules — Participants will receive oral administration of TJ0113.
  Arms: Food Effect: 200 mg C1: fasting-fed; Food Effect: 200 mg C2: fed-fasting; Multiple Ascending Dose (MAD): 200 mg QD; Multiple Ascending Dose (MAD): 300 mg BID; Multiple Ascending Dose (MAD): 400 mg QD; Single Ascending Dose (SAD): 160 mg; Single Ascending Dose (SAD): 260 mg; Single Ascending Dose (SAD): 400 mg; Single Ascending Dose (SAD): 540 mg; Single Ascending Dose (SAD): 720 mg; Single Ascending Dose (SAD): 80 mg
Other: Placebo — Participants will receive oral administration of Placebo.
  Arms: Multiple Ascending Dose (MAD): placebo; Single Ascending Dose (SAD): placebo

SUMMARY:
The study included three clinical studies, namely a single ascending dose (SAD) study, a multiple ascending dose (MAD) study, and a high-fat diet food effect (FE) study.

DETAILED DESCRIPTION:
Study 1: SAD study A single-center, randomized, double-blind, placebo-controlled, single ascending dose study of TJ0113 capsules in healthy subjects. Six dose groups (A1-A6) were established, with doses of 80 mg, 160 mg, 260 mg, 400 mg, 540 mg, and 720 mg, respectively.

A total of 72 healthy adult subjects (12 per group) were enrolled, including both males and females. Subjects in each dose group were randomized in a 5:1 ratio to receive either the investigational product, TJ0113 capsules, or placebo (10 subjects received the investigational product and 2 subjects received placebo). Two subjects in the 80 mg dose group were set as a sentinel arm and were randomized in a 1:1 ratio to receive either TJ0113 capsules or placebo. After completing the 24-hour safety observation following sentinel dosing, the remaining 10 subjects in the 80 mg dose group were randomized in a 9:1 ratio to receive either TJ0113 capsules or placebo.

Study 2: MAD study In the single-center, randomized, double-blind, placebo-controlled, MAD study of TJ0113 capsules in healthy subjects, 3 dose groups (B1 to B3) of 200 mg once daily(QD), 400 mg QD, 300 mg twice daily(BID )were set.

A total of 36 healthy adult subjects (12 per group) were enrolled, including both males and females. Subjects in each dose group were randomized in a 5:1 ratio to receive either the investigational product, TJ0113 capsules, or placebo (10 subjects received the investigational product and 2 subjects received placebo). Subjects in the 200 mg and 400 mg dose groups received once-daily (QD) dosing, while subjects in the 300 mg BID dose group received twice-daily (BID) dosing administered with warm water, for 7 consecutive days (only one dose in the morning on Day 7).

Study 3: FE study A single-center, single-dose, randomized, open-label, 2-sequence, 2-period, crossover study to evaluate the effect of a standard high-fat diet on the pharmacokinetics of TJ0113 capsules after single oral administration (200 mg) in healthy subjects.

A total of 20 healthy adult subjects were enrolled in this period and randomized in a 1:1 ratio to 2 dosing sequences (C1: fasting-fed; C2: fed-fasting), with 10 subjects per group (all receiving the investigational product TJ0113 capsule). Each dosing sequence consisted of 2 cycles with 1 dose administered in each cycle. Group C1 received the dose in a fasting state during the first cycle and in a fed state during the second cycle; Group C2 received the dose in a fed state during the first cycle and in a fasting state during the second cycle . The two cycles were separated by a 7-day washout period.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate in the clinical trial, sign the informed consent form, understand and agree to follow the protocol, have a full understanding of trial contents, process, and possible adverse reactions, and indicate the date of signing;
2. Aged 18 ~ 55 years (inclusive), Chinese healthy male or female;
3. Body weight ≥ 50 kg (male) or ≥ 45 kg (female), body mass index (BMI) within the range of 19.0 ~ 26.0 kg/m2 (inclusive);
4. Subjects and their partners have no plans for pregnancy, donation of sperm or eggs, and voluntarily take effective contraceptive measures (such as abstinence, condom, etc.) from the screening phase until 6 months after the end of the trial;
5. Able to communicate well with the investigator, understand and agree to follow all requirements of this trial.

Exclusion Criteria:

1. Subjects with a history or current presence of chronic diseases involving the cardiovascular, respiratory, urinary, nervous, psychiatric, hematological, endocrine and metabolic (diabetes, thyroid disease, adrenal disease), and immune systems, and deemed unsuitable for participation by the investigator.
2. Subjects who have received surgery within 3 months before screening, or plan to receive surgery during the trial; or have received medical or surgical treatment (such as gastrointestinal surgery) permanently changing the absorption, distribution, metabolism and excretion of oral drugs (except for hernia repair); a history of abdominal surgery, such as cholecystectomy (except for uncomplicated appendectomy and endoscopic treatment of gastrointestinal polyps after 6 months);
3. Subjects with dysphagia or gastrointestinal, liver, or kidney diseases (regardless of whether they have been cured) within 6 months before screening that could affect drug absorption or excretion;
4. History of clinically significant drug allergy or specific allergic diseases (such as asthma, urticaria) or known hypersensitivity to the investigational product or its excipients;
5. Subjects who have used any drugs (including prescription drugs, over-the-counter drugs, Chinese herbal medicines, etc.) or supplements within 14 days before the first dose;
6. Subjects with abnormal and clinically significant results on physical examination, vital signs, laboratory tests (blood routine test, urinalysis + specific gravity, blood biochemistry, coagulation function, etc.) at screening and baseline;
7. Subjects with clinically significant 12-lead ECG abnormalities at screening or baseline, or with an average QTcF (corrected QT interval using Fridericia's formula) >450 ms for males, >470 ms for females, QRS >120 ms, or a history of long QT syndrome.
8. Subjects who have special dietary requirements and cannot abide by the standard diet;
9. Subjects who are difficult to collect blood samples or cannot tolerate venipuncture, and have a history of fainting at the sight of blood or needles;
10. Subjects who have blood donation or non-physiological blood loss ≥ 400 mL (including trauma, blood collection, blood donation, etc., except for physiological blood loss in females) within 3 months before screening, or blood transfusion; or blood donation or non-physiological blood loss ≥ 200 mL within 1 month before screening; or blood donation or blood components planned during the study or within 3 months after the end of the study;
11. Subjects who have excessively used nicotine products (more than 5 cigarettes in average daily) within 3 months before screening and cannot stop using any tobacco products throughout the trial; subjects with positive urine cotinine tests;
12. Subjects who have consumed more than 14 units of alcohol per week within 6 months prior to screening (1 unit of alcohol ≈ 360 mL of beer or 45 mL of 40% alcohol spirits or 150 mL of wine), have a positive alcohol breath test at baseline (breath alcohol content >0.0 mg/100 mL), or cannot abstain from alcohol during the trial;
13. Subjects who have long-term excessive consumption of tea, coffee, or caffeinated beverages (more than 8 cups per day, 1 cup = 200 mL) within the year prior to screening; subjects who have consumed any foods or beverages containing caffeine, alcohol, xanthine, or grapefruit components, or other substances that affect drug absorption, distribution, metabolism, and excretion (such as coffee, tea, chocolate, etc.) within 48 hours before the first dose;
14. Subjects who have received live vaccine inoculations within 14 days before screening or plan to receive them during the trial or within 1 month after dosing, including but not limited to measles, mumps, rubella, varicella, yellow fever, rabies, Bacillus Calmette-Guerin Vaccine (BCG), typhoid vaccine, COVID-19 vaccine, etc.;
15. Subjects who have febrile illness or active infection within 14 days before screening;
16. Subjects who have used any known hepatic enzyme inducers or inhibitors within 30 days before the first dose;
17. Subjects with drug addiction or positive drug abuse tests, or a history of drug abuse/dependence or drug use within 1 year before screening;
18. Subjects with positive results on infectious disease screening, including positive human immunodeficiency virus (HIV) antigen/antibody, positive hepatitis B surface antigen (HBsAg) quantification, positive hepatitis C virus (HCV) antibody, positive Treponema pallidum antibody tests;
19. Subjects with positive pregnancy tests at screening or baseline, who are pregnant, breastfeeding, or planning to become pregnant during the trial, or men or women of childbearing potential who are unwilling to use effective contraception for 6 months after the last dose;
20. Subjects who are unable to comply with all requirements of the study or still need to engage in or plan to participate in strenuous physical activity or exercise during the trial, including body contact or collision sports;
21. Subjects who have participated in other clinical trials of drugs or medical devices within 3 months before screening, and received investigational products or medical devices; or planned to participate in other trials during the study period; or within 5 half-lives of another drug before screening (if 5 half-lives exceed 3 months);
22. Employees or related personnel of the investigator, study site, sponsor, or contract research organization (CRO).Subjects who have other conditions that could impact compliance in the opinion of the investigator or who are unable to participate in the trial due to personal reasons.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 130 (Actual)
Dates: Start 2023-08-04 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2024-04-03 (Actual)

PRIMARY OUTCOMES:
Treatment-emergent adverse event (TEAE) incidence of TJ0113 capsules after single oral administration in SAD study | Within 12 days after the last administration
  Types, incidence rates, and severity of adverse events. Safety evaluation indicators include, but are not limited to, the following items: adverse events, physical examination, vital signs, electrocardiogram (ECG), laboratory test results (coagulation function, complete blood count, blood biochemistry, urinalysis plus urine specific gravity, etc.)
Treatment-emergent adverse event (TEAE) incidence of TJ0113 capsules after multiple oral administration in MAD study | Within 12 days after the last administration
  Types, incidence rates, and severity of adverse events. Safety evaluation indicators include, but are not limited to, the following items: adverse events, physical examination, vital signs, electrocardiogram (ECG), laboratory test results (coagulation function, complete blood count, blood biochemistry, urinalysis plus urine specific gravity, etc.)

SECONDARY OUTCOMES:
Maximum concentration (Cmax) of TJ0113 capsules after oral administration in SAD study | Within 72 hours after the last administration
  PK parameters for the SAD study mainly included maximum concentration (Cmax)
Area under the plasma concentration versus time curve (AUC) of TJ0113 capsules after oral administration in SAD study | Within 72 hours after the last administration
  PK parameters for the SAD study mainly included area under the plasma concentration versus time curve (AUC)
Half life（t1/2） of TJ0113 capsules after oral administration in SAD study | Within 72 hours after the last administration
  PK parameters for the food effect study mainly included half life（t1/2）
Time to maximum concentration (Tmax) of TJ0113 capsules after oral administration in SAD study | Within 72 hours after the last administration
  PK parameters for the food effect study mainly included time to maximum
Maximum concentration (Cmax) of TJ0113 capsules after oral administration in MAD study | Within 72 hours after the last administration
  PK parameters for the MAD study mainly included maximum concentration (Cmax)
Area under the plasma concentration versus time curve (AUC) of TJ0113 capsules after oral administration in MAD study | Within 72 hours after the last administration
  PK parameters for the MAD study mainly included area under the plasma concentration versus time curve (AUC)
Half life（t1/2） of TJ0113 capsules after oral administration in MAD study | Within 72 hours after the last administration
  PK parameters for the food effect study mainly included half life（t1/2）
Time to maximum concentration (Tmax) of TJ0113 capsules after oral administration in MAD study | Within 72 hours after the last administration
  PK parameters for the food effect study mainly included time to maximum
Maximum concentration (Cmax) of TJ0113 capsules after oral administration with a standard high-fat diet in FE | Within 72 hours after the last administration
  PK parameters for the FE study mainly included maximum concentration (Cmax)
Area under the plasma concentration versus time curve (AUC) of TJ0113 capsules after oral administration with a standard high-fat diet in FE study | Within 72 hours after the last administration
  PK parameters for the FE study mainly included area under the plasma concentration versus time curve (AUC)
Half life（t1/2） of TJ0113 capsules after oral administration with a standard high-fat diet in FE study | Within 72 hours after the last administration
  PK parameters for the food effect study mainly included half life（t1/2）
Time to maximum concentration (Tmax) of TJ0113 capsules after oral administration with a standard high-fat diet in FE study | Within 72 hours after the last administration
  PK parameters for the food effect study mainly included time to maximum
Treatment-emergent adverse event (TEAE) incidence of TJ0113 capsules after multiple oral administration with a standard high-fat diet in FE study | Within 15 days after the last administration
  Types, incidence rates, and severity of adverse events. Safety evaluation indicators include, but are not limited to, the following items: adverse events, physical examination, vital signs, electrocardiogram (ECG), laboratory test results (coagulation function, complete blood count, blood biochemistry, urinalysis plus urine specific gravity, etc.)

CONTACTS AND LOCATIONS:
Overall Officials: Jian Chen, Principal Investigator — Zhejiang Hospital
Locations (1):
- Zhejiang Xiaoshan hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No